CLINICAL TRIAL: NCT01250210
Title: Evaluation of Pharmacodynamic Effects on Ovulation Suppression and Cycle Control of Three Agile Contraceptive Patches Containing Different Doses of Ethinyl Estradiol(EE)During Three Cycles of Administration
Brief Title: Evaluation of Pharmacodynamic Effects on Ovulation and Cycle Control
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agile Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATI-CL11
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Ovulation Suppression
Keywords: contraception; pregnancy prevention
MeSH Terms: interventions — ethinyl estradiol, levonorgestrel drug combination; Contraception; Hormonal Contraception; Administration, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- AG200-15 (Experimental): Drug intervention with levonorgestrel and ethinyl estradiol : AG200-15 a transdermal contraceptive system containing 2.60 mg of levonorgestrel and 2.30 mg of ethinyl estradiol.
  Interventions: Drug: levonorgestrel and ethinyl estradiol
- AG200 (Experimental): Drug intervention with levonorgestrel and ethinyl estradiol: AG200 a transdermal contraceptive system containing 2.17 mg of levonorgestrel and 1.92 of ethinyl estradiol.
  Interventions: Drug: levonorgestrel and ethinyl estradiol
- AG200LE (Experimental): Drug intervention with levonorgestrel and ethinyl estradiol: AG200LE a transdermal contraceptive system containing 2.17 mg of levonorgestrel and 1.28 mg of ethinyl estradiol.
  Interventions: Drug: levonorgestrel and ethinyl estradiol

INTERVENTIONS:
Drug: levonorgestrel and ethinyl estradiol — pregnancy prevention
  Other Names: contraception; hormonal contraception; transdermal

SUMMARY:
Evaluate the adequacy of ovulation suppression, cycle control, and safety of three transdermal contraceptive delivery systems (TCDSs).

DETAILED DESCRIPTION:
The primary objective was to evaluate the adequacy of ovulation suppression, cycle control, and safety of three transdermal contraceptive delivery systems (TCDSs) containing 2 different doses of levonorgestrel (LNG) and 3 different doses of ethinyl estradiol (EE) during 3 consecutive cycles of administration of each treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult women, ages 18-45.
2. Cycles with a usual duration between 21 and 35 days and an individual variation of +/ 3 days.
3. Normotensive (blood pressure < 140/90 mm Hg at rest) at screening and randomization visits (Visits 1 and 2).
4. Willing to use a non-hormonal method of contraception for the entire duration of the study, or
5. Have already undergone previous bilateral tubal ligation OR vasectomized partner OR not at risk of pregnancy.
6. Willing to refrain from excessive use of alcohol during the entire duration of the study.
7. Willing to give informed consent to participate in the study.

Exclusion Criteria:

1. History of significant medical illness or seizures.
2. Positive hepatitis B or C antibody or positive human immunodeficiency virus (HIV) antibody.
3. Known or suspected pregnancy.
4. A recent abnormal cervical smear - low-grade squamous intraepithelial lesion (SIL) or higher in the Bethesda System - which has not been resolved or treated.
5. Any disorder that contraindicates the use of contraceptive steroids i.e., history of heart attack and stroke, blood clots in the legs, lungs or eyes, history of blood clots in the deep veins of the legs, known or suspected breast cancer, hepatitis or yellowing of the whites of the eyes or the skin (jaundice) during pregnancy or during previous use of hormonal contraceptives, headaches with neurological symptoms, disease of heart valves with complications.
6. Uncontrolled thyroid disorder.
7. History of or existing thromboembolic disorder, vascular disease, cerebral vascular, or coronary artery disease.
8. Undiagnosed abnormal genital bleeding.
9. Known or suspected breast carcinoma, endometrial carcinoma, or estrogen-dependent neoplasia.
10. History or presence of dermal hypersensitivity in response to topical application.
11. Use of an injectable hormonal contraceptive (e.g. Depo-Provera®) within 6 months prior to Day 1.
12. Use of a contraceptive implant (e.g. Implanon® or Jadelle®) or hormone-medicated intrauterine device within 2 months (60 days) prior to Day 1.
13. Use of OCs or other sex steroid hormones within 60 days prior to Day 1.
14. Women who are breast-feeding or are within 2 months of stopping breast-feeding.
15. Status post-partum or post-abortion within a period of 2 months prior to Day 1.
16. Chronic use of any medication that might interfere with the metabolism of hormone contraceptives (e.g., rifampin, barbiturates, phenytoin, primidone, topiramate, carbamazepine, phenylbutazone, ritonavir, modafinil, St John's Wort etc.) or use within the past 3 months prior to Day 1.
17. Administration of investigational drug within 30 days prior to Day 1.
18. A history (within prior 12 months) of drug or alcohol abuse.
19. Women who smoke more than 4-5 cigarettes daily.
20. History of skin sensitivity to adhesives.
21. Use of over-the-counter medications or herbals that might interfere with the metabolism of hormone contraceptives within 3 days prior to wearing the first patch.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Garner, MD, MPH, Study Director — Agile Therapeutics
Locations (11):
- United States (11):
  - Tucson, Arizona
  - San Diego, California
  - Denver, Colorado
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Sandy Springs, Georgia
  - Cary, North Carolina
  - Winston-Salem, North Carolina
  - Jenkintown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Bristol, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned enrollment included: approximately 30 subjects in the AG200LE treatment group, 30 subjects in the AG200 treatment group and 20 to 30 subjects in the AG200 15 treatment group. Actual enrollment included: 45 subjects in the AG200 treatment group; 45 subjects in the AG200LE treatment group; and 33 subjects in the AG200-15 treatment group.
Pre-assignment Details: : Subjects enrolled were healthy adult women aged 18-45 years with a history of regular menstrual cycles (i.e., lasting between 21 and 35 days) and no disorders precluding hormonal contraceptive use.
Groups:
- AG200LE Transdermal Contraceptive Delivery System: a 12.5 cm2 patch (Lot #27621) containing 2.17 LNG/1.28 EE mg (designed to deliver approximately: 0.075 LNG/0.015 EE mg/day).
- AG200 Transdermal Contraceptive Delivery System: a 12.5 cm2 patch (Lot #27620) containing 2.17 LNG/1.92 EE mg (designed to deliver approximately: 0.1 LNG/0.02 EE mg/day).
- AG200-15 Transdermal Contraceptive System: a 15 cm2 patch (Lot #27620) containing 2.60 LNG/2.30 EE mg (designed to deliver approximately: 0.12 LNG/0.025 EE mg/day).
Period: Overall Study
Arm/Group | AG200LE Transdermal Contraceptive Delivery System | AG200 Transdermal Contraceptive Delivery System | AG200-15 Transdermal Contraceptive System
Started (Number of participants enrolled.) | 45 | 45 | 33
Completed | 41 | 41 | 25
Not Completed | 4 | 4 | 8

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | AG200LE Transdermal Contraceptive Delivery System | AG200 Transdermal Contraceptive Delivery System | AG200-15 Transdermal Contraceptive System | Total
Number analyzed (Participants) | 43 | 44 | 31 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 43 | 44 | 31 | 118
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (7.4) | 31 (6.9) | 32.1 (7.8) | 31.6 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 44 | 31 | 118
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 44 | 31 | 118

OUTCOME MEASURES:

1. Primary Outcome: Ovulation Suppression in Three Treatment Groups Over 3 Cycles
Description: Ovulation suppression measured by possible ovulation. Possible ovulation is defined as cycles with greatest progesterone level ≥4.7 ng/mL across Cycles 1-3 combined for each Arm/Group. The following four primary analysis datasets are:
  Intent-to-treat (ITT): At least 1 study patch was applied and at least 1 progesterone measurement is available at 1 of the nominal data collection points.
  Complete progesterone: At least 1 study patch was applied and at least 3 progesterone measurements are available across any of the data collection points.
  Perfect compliance: If no patch has been off >1 day and no more than 1 day has elapsed between patch changes.
  Verifiable compliance: is a cycle during which at least 1 study patch was applied and where LNG and EE measurements were available at each of the nominal data collection points of Days 8, 15, and 22, and all values were above the lower detection limit.
Time Frame: 3 months
Population: ITT, perfect compliance, complete progesterone, verifiable compliance
Measure: Number; unit: %of cycles with possible ovulation
Units Other Than Participants: Total number of cycles
Groups:
- AG200LE: a 12.5 cm2 patch (Lot #27621) containing 2.17 LNG/1.28 EE mg (designed to deliver approximately: 0.075 LNG/0.015 EE mg/day).
- AG200: a 12.5 cm2 patch (Lot #27620) containing 2.17 LNG/1.92 EE mg (designed to deliver approximately: 0.1 LNG/0.02 EE mg/day).
- AG200-15: a 15 cm2 patch (Lot #27620) containing 2.60 LNG/2.30 EE mg (designed to deliver approximately: 0.12 LNG/0.025 EE mg/day).
Arm/Group | AG200LE | AG200 | AG200-15
Number analyzed (Participants) | 35 | 32 | 23
Number analyzed (Total number of cycles) | 104 | 92 | 61
%of cycles with possible ovulation
  ITT, perfect compliance | 36.5 | 20.7 | 11.5
  Complete progesterone, perfect compliance | 36.9 | 20.7 | 11.7
  ITT, verifiable compliance | 32.5 | 14.9 | 12.0
  Complete progesterone, verifiable compliance | 32.5 | 14.9 | 12.0

2. Primary Outcome: Cycle Control
Description: The incidence of breakthrough bleeding (BTB) and/or spotting (S) episodes in Cycle 3 for ITT cycles. A BTB/S episode was defined as any number of days with BTB and/or BTS preceded and followed by at least 2 bleeding-free days.
Time Frame: 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | AG200LE | AG200 | AG200-15
Number analyzed (Participants) | 42 | 42 | 27
number of episodes | 0.29 (0.46) | 0.29 (0.46) | 0.15 (0.36)

ADVERSE EVENTS:
Description: Adverse Events were analyzed for the Safety population. Adverse Events analyzed are based on Organ System class only.
Arm/Group | AG200LE | AG200 | AG200-15
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/44 | 0/31
Other Adverse Events (participants affected / at risk) | 19/43 | 29/44 | 19/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG200LE (N=43) | AG200 (N=44) | AG200-15 (N=31)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) | 6 (6) | 5 (5)
General disorders and administration site conditions (General disorders) | 2 (2) | 5 (5) | 5 (5)
Immune system disorders (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Infections and infestations (Infections and infestations) | 4 (4) | 2 (2) | 6 (6)
Investigations (Investigations) | 2 (2) | 3 (3) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (1) | 5 (5) | 3 (3)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 3 (3) | 6 (6) | 6 (6)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | 4 (4)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6) | 6 (6)
Vascular disorders (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications must be reviewed and approved by sponsor